CLINICAL TRIAL: NCT03377452
Title: Diagnosis and Treatment of Sleep Apnea in Women Veterans
Brief Title: Treating Sleep Apnea in Women Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIR 16-244
Record Dates: First submitted 2017-12-14; First posted 2017-12-19 (Actual); Results first posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-01

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: Individuals will be assigned to one of two programs simultaneously
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors will be blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acceptance and the Behavioral Changes to Treat Sleep Apnea (ABC-SA) (Experimental): Six session manual-based program using acceptance-and commitment therapy (ACT) framework, behavior change strategies and sleep apnea/PAP education. Sessions delivered in individual format, either in-person or via telehealth.
  Interventions: Behavioral: Acceptance and the Behavioral Changes to Treat Sleep Apnea (ACB-SA)
- Non-directive sleep apnea education control (Active Comparator): Six session sleep apnea and PAP education program. Sessions delivered in individual format, either in-person or via telehealth.
  Interventions: Behavioral: Non-directive sleep apnea education control

INTERVENTIONS:
Behavioral: Acceptance and the Behavioral Changes to Treat Sleep Apnea (ACB-SA) — Six session manual-based program using acceptance-and commitment therapy (ACT) framework, behavior change strategies and sleep apnea/PAP education. Sessions delivered in individual format, either in-person or via telehealth.
  Arms: Acceptance and the Behavioral Changes to Treat Sleep Apnea (ABC-SA)
Behavioral: Non-directive sleep apnea education control — Six session sleep apnea and PAP education program. Sessions delivered in individual format, either in-person or via telehealth.
  Arms: Non-directive sleep apnea education control

SUMMARY:
This study is a randomized controlled trial (RCT) to test two sleep apnea education programs for women Veterans newly diagnosed with sleep apnea (SA) who are prescribed positive airway pressure (PAP) therapy. This education program is designed to improve participants' sleep quality and help them to adjust to PAP therapy.

Participants undergo a sleep and health assessment that is performed prior to beginning the education program. This assessment includes wearing a wrist actigraph to measure sleep and wake periods for 7 days and nights, and answering questionnaires about sleep habits and health. Participants are randomly assigned to one of two 6-week programs (intervention or educational control) provided by a study interventionist. Follow-up sleep and health assessments will be conducted at the end of the 6-week program and 3-months later. PAP usage data will be collected remotely for 6-months from PAP therapy initiation.

DETAILED DESCRIPTION:
Sleep disordered breathing (SDB) is associated with significant adverse health consequences including cardiovascular disease, motor vehicle accidents, daytime functional impairments and mortality risk. Although SDB is more common among men than women, it still impacts 17% of women in the general population. [The investigators' preliminary evidence suggests it is even more common among women Veterans who receive VA care.] The recommended first-line therapy for most patients with SDB is positive airway pressure therapy (PAP). Published studies show that women have lower PAP adherence than men, particularly in the US, yet the investigators are not aware of data comparing men and women Veterans. Because women Veterans experience significant sleep disturbance and other consequences of sleep disorders, adjusting to PAP therapy may be quite difficult. To date, studies have not tested interventions specifically designed to improve PAP adherence among women, accounting for important sleep-related and social factors.

This study is a randomized controlled trial (RCT) to test the efficacy of a program combining patient education with behavioral techniques and exercises from acceptance and commitment therapy (ACT) to improve adherence to PAP therapy. Women Veterans 18 years and older, who have received care at the VA Greater Los Angeles Healthcare System, and who have at least 1 risk factor for SDB will be recruited for this study. Screening for sleep apnea will be performed in the participant's home using a WatchPAT device. Both objective (actigraphy) and self-report (questionnaire/diary) sleep measures will be collected, as well as other health-related measures. Participants with an Apnea-Hypopnea Index (AHI) of 5 or higher, and who meet all inclusion/exclusion criteria will be randomized to one of two programs: Acceptance and the Behavioral Changes to Treatment of Sleep Apnea (ABC-SA) or a non-directive sleep apnea education control.

PAP devices, along with education about SDB and sleep, will be provided to participants as part of the 6-session intervention and control programs. Follow-up assessments will be conducted immediately following the intervention/control and after 3-months.

Main study outcomes (sleep quality and PAP adherence) will be assessed 3 months after PAP initiation, and PAP adherence will be tracked remotely for 6 months. Data will be analyzed using "intention to treat" principles, using appropriate statistical methods for clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling women Veterans aged 18 years and older
* Received care from a Veterans Health Administration (VHA) facility
* Have a least one risk factor for sleep apnea (e.g., hypertension, obesity, or age 50 years or older)
* Diagnosed as having sleep apnea with an AHI of 5 or greater

Exclusion Criteria:

* Currently using a treatment for sleep apnea
* Current pregnancy
* Active substance user or in recovery with < 90 days of sobriety
* Too ill to engage in study procedures
* Do not have transportation to the medical center
* Unable to self-consent (e.g., due to cognitive impairment)
* Unstable housing
* Does not have sleep apnea
* Another sleep disorder (e.g., restless legs syndrome, circadian rhythm sleep disorder) accounts for sleep disturbance
* No sleep complaints or symptoms

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is for women Veterans.
Enrollment: 90 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Martin, PhD, Principal Investigator — VA Greater Los Angeles Healthcare System, Sepulveda, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, Sepulveda, CA, Sepulveda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Moghtaderi I, Kelly MR, Carlson GC, Fung CH, Josephson KR, Song Y, Swistun D, Zhu R, Mitchell M, Lee D, Badr MS, Washington DL, Yano EM, Alessi CA, Zeidler MR, Martin JL. Identifying gaps in clinical evaluation and treatment of sleep-disordered breathing in women veterans. Sleep Breath. 2023 Oct;27(5):1929-1933. doi: 10.1007/s11325-022-02765-1. Epub 2022 Dec 16. PMID 36525174
- [Result] Saldana KS, McGowan SK, Martin JL. Acceptance and Commitment Therapy as an Adjunct or Alternative Treatment to Cognitive Behavioral Therapy for Insomnia. Sleep Med Clin. 2023 Mar;18(1):73-83. doi: 10.1016/j.jsmc.2022.09.003. PMID 36764788
- [Result] Carlson GC, Kelly MR, Grinberg AM, Mitchell M, McGowan SK, Culver NC, Kay M, Alessi CA, Washington DL, Yano EM, Martin JL. Insomnia Precipitating Events among Women Veterans: The Impact of Traumatic and Nontraumatic Events on Sleep and Mental Health Symptoms. Behav Sleep Med. 2021 Sep-Oct;19(5):672-688. doi: 10.1080/15402002.2020.1846537. Epub 2020 Nov 30. PMID 33251855
- [Result] Carlson GC, Kelly MR, Mitchell M, Josephson KR, McGowan SK, Culver NC, Kay M, Alessi CA, Fung CH, Washington DL, Hamilton A, Yano EM, Martin JL. Benefits of Cognitive Behavioral Therapy for Insomnia for Women Veterans with and without Probable Post-Traumatic Stress Disorder. Womens Health Issues. 2022 Mar-Apr;32(2):194-202. doi: 10.1016/j.whi.2021.10.007. Epub 2021 Nov 21. PMID 34815139
- [Result] Saldana KS, Carlson GC, Revolorio K, Kelly MR, Josephson KR, Mitchell MN, Culver N, Kay M, McGowan SK, Song Y, Deleeuw C, Martin JL. Values Expressed by Women Veterans Receiving Treatment for Chronic Insomnia Disorder. Behav Sleep Med. 2024 May-Jun;22(3):340-352. doi: 10.1080/15402002.2023.2260517. Epub 2023 Sep 25. PMID 37749876
- [Result] Ravyts SG, Erickson AJ, Washington DL, Yano EM, Carlson GC, Mitchell MN, Kelly M, Alessi CA, McGowan SK, Song Y, Martin JL, Dzierzewski JM. A non-inferiority randomized controlled trial comparing behavioral sleep interventions in women veterans: An examination of pain outcomes. J Psychosom Res. 2023 Dec;175:111536. doi: 10.1016/j.jpsychores.2023.111536. Epub 2023 Oct 21. PMID 37913677

RESULTS

PARTICIPANT FLOW:
Groups:
- Acceptance and the Behavioral Changes to Treat Sleep Apnea (ABC-SA): Six session manual-based program using acceptance and commitment therapy (ACT) framework, behavior change strategies and sleep apnea/PAP education.
  Sessions delivered in individual format, either in-person or via telehealth.
Period: Overall Study
Arm/Group | Acceptance and the Behavioral Changes to Treat Sleep Apnea (ABC-SA) | Non-directive Sleep Apnea Education Control
Started | 44 | 46
Post Treatment | 40 | 44
3 Month Follow-up | 39 | 40
Completed | 39 | 40
Not Completed | 5 | 6
Not completed — Refused assessment | 0 | 2
Not completed — Lost to Follow-up | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acceptance and the Behavioral Changes to Treat Sleep Apnea (ABC-SA) | Non-directive Sleep Apnea Education Control | Total
Number analyzed (Participants) | 44 | 46 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (13.2) | 52.7 (12.6) | 53.2 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 46 | 90
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 14 | 25
  Not Hispanic or Latino | 33 | 32 | 65
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 14 | 10 | 24
  White | 27 | 27 | 54
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 0 | 2 | 2
Sleep Quality [Mean (Standard Deviation); unit: units on a scale] — Total score on the Pittsburgh Sleep Quality Index. Scores range from 0 to 21. Higher scores indicate worse outcome.
  units on a scale | 9.4 (4.1) | 9.1 (4.3) | 9.3 (4.2)
Baseline AHI [Mean (Standard Deviation); unit: mean events per hour] — Apnea-Hypopnea Index (AHI) was calculated from overnight monitoring with a WatchPat 200 device. The AHI is the average number of apneas and hypopneas that occur per hour of sleep during the recording. An AHI > 5 is considered positive for sleep apnea. As AHI increases, the severity of sleep apnea increases.
  mean events per hour | 23.3 (15.4) | 20.5 (12.0) | 21.9 (13.8)
Insomnia Severity Index [Mean (Standard Deviation); unit: units on a scale] — Total Score on Insomnia Severity Index. Total score ranges from 0-28 where higher scores indicate worse outcome.
  units on a scale | 15.4 (5.7) | 12.7 (6.3) | 14.0 (6.1)

OUTCOME MEASURES:

1. Primary Outcome: PAP Adherence
Description: Number of nights positive airway pressure (PAP) was used >=4 hours during the first 90 days measured by remote monitoring. Number of nights range from 0 to 90 nights. More nights indicate better outcome. Remote monitoring data were available for all participants even if lost to follow-up for other measures. The sample size for this outcome is larger than for other outcomes as a result.
Time Frame: Three months after PAP initiation
Measure: Mean (Standard Error); unit: Number of nights
Arm/Group | Acceptance and the Behavioral Changes to Treat Sleep Apnea (ABC-SA) | Non-directive Sleep Apnea Education Control
Number analyzed (Participants) | 44 | 46
Number of nights | 32.9 (4.49) | 25.67 (4.03)
Statistical Analysis 1: Comparison: Acceptance and the Behavioral Changes to Treat Sleep Apnea (ABC-SA) vs Non-directive Sleep Apnea Education Control; Test type: Superiority; p = 0.2313, t-test, 2 sided; Mean Difference (Final Values) = 7.26, 95% CI 2-sided [-4.71 to 19.22], Standard Error of Mean 6.02

2. Primary Outcome: Sleep Quality by Patient-reported Sleep Questionnaire
Description: Self-reported sleep quality assessed with a brief patient questionnaire assessing multiple aspects of sleep quality.
  Total score on the Pittsburgh Sleep Quality Index will be used as a measure of sleep quality. Scores range from 0 to 21. Higher scores indicate worse outcome. This measure is available only for participants who were not lost to follow-up.
Time Frame: Baseline, Three months from the date of the last intervention/control session (typically 12-16 weeks after the final session)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Acceptance and the Behavioral Changes to Treat Sleep Apnea (ABC-SA) | Non-directive Sleep Apnea Education Control
Number analyzed (Participants) | 39 | 40
score on a scale
  Baseline | 9.41 (0.63) | 9.11 (0.61)
  Three months from the date of the last intervention/control session | 6.37 (0.59) | 9.39 (0.58)
Statistical Analysis 1: Comparison: Acceptance and the Behavioral Changes to Treat Sleep Apnea (ABC-SA) vs Non-directive Sleep Apnea Education Control; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -3.31, 95% CI 2-sided [-4.91 to -1.72], Standard Error of Mean 0.81 — The parameter estimate is the change in the outcome from baseline to 3-months after the last intervention/control session for the intervention group versus the same change in the control group

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from enrollment and through the end of the 3-month follow-up period.
Description: Does not differ from ClinicalTrials.gov definitions.
Arm/Group | Acceptance and the Behavioral Changes to Treat Sleep Apnea (ABC-SA) | Non-directive Sleep Apnea Education Control
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/46
Other Adverse Events (participants affected / at risk) | 0/44 | 0/46

LIMITATIONS AND CAVEATS:
The study transitioned from in-person to telehealth visits during the COVID-19 pandemic. As a result, actigraphy could not be collected from some participants and the target sample size was not achieved for this secondary outcome. PAP devices used in the trial were recalled by the manufacturer during the final year of enrollment. Impacted participants were contacted and provided assistance. PAP devices from a different manufacturer were purchased for remaining participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-24): https://cdn.clinicaltrials.gov/large-docs/52/NCT03377452/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-24): https://cdn.clinicaltrials.gov/large-docs/52/NCT03377452/ICF_001.pdf